CLINICAL TRIAL: NCT03018444
Title: The Effect of HMG-CoA Reductase Inhibition on Postprandial GLP-1 Secretion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Responsible Party: Principal Investigator, Filip Krag Knop, Professor, University Hospital, Gentofte, Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: H-16034243
Record Dates: First submitted 2017-01-10; First posted 2017-01-12 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-03

CONDITIONS: Diabetes Mellitus, Type 2; Hydroxymethylglutaryl-CoA Reductase Inhibitors
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- Atorvastatin (Experimental): 2 weeks treatment with Atorvastatin (1st week 40 mg once daily on day, 2nd week 80 mg (2x40mg) once daily)
  Interventions: Drug: Atorvastatin
- Placebo (Placebo Comparator): 2 weeks treatment with placebo tablets of comparable sizes and color to the Atorvastatin tablets (1st week one tablet once daily, 2nd week two tablets once daily)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Atorvastatin — Atorvastatin tablet
  Arms: Atorvastatin
Other: Placebo — Placebo tablet
  Arms: Placebo

SUMMARY:
The primary objective of the present study is to evaluate the effect of HMG-CoA reductase inhibition during 14 days on the postprandial plasma GLP-1 response in healthy individuals. Secondary objectives include the evaluation of HMG-CoA reductase inhibition on postprandial glucose tolerance, gallbladder emptying, gastric emptying, plasma responses of lipids, bile acids and pancreatic and enteric hormones known to influence glucose metabolism and appetite, and faecal content of bile acids and gut microbiota composition.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) >18.5 kg/m2 and <35 kg/m2
* Caucasian ethnicity
* Normal haemoglobin
* Glycated haemoglobin (HbA1c) <43 mmol/mol
* Fasting plasma glucose <6 mmol/l
* Informed and written consent

Exclusion Criteria:

* Diabetes
* First-degree relatives with diabetes (both type 1 diabetes and type 2 diabetes)
* Liver disease (serum alanine aminotransferase (ALAT) and/or serum aspartate aminotransferase (ASAT) >2 times normal values) or history of hepatobiliary disorder
* Gastrointestinal disease, previous intestinal resection, cholecystectomy or any major intra-abdominal surgery
* Reduced kidney function or nephropathy (estimated glomerular filtration rate (eGFR) <60 ml/min/1.73 m2 (based on serum creatinine) and/or albuminuria
* Taking any kind of medicine on a regular basis
* Intake of antibiotics two months prior to study
* Active or recent malignant disease
* Any treatment or condition requiring acute or sub-acute medical or surgical intervention
* Any condition considered incompatible with participation by the investigators
* If the subjects receive any antibiotic treatment while included in the study they will be excluded

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-10; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Postprandial GLP-1 secretion | 240 min

SECONDARY OUTCOMES:
Postprandial Bile Acid Composition | 240 min
Postprandial total plasma Bile Acid | 240 min
Postprandial Glucose Tolerance | 240 min
Postprandial plasma lipid response | 240 min
Postprandial GIP secretion | 240 min
Enteric hormones known to influence glucose metabolism | 240 min
Gallbladder emptying | 240 min
Faecal content of bile acid | One sample collected on day 12 or 13 of the intervention
Gut microbiota composition | One sample collected on day 12 or 13 of the intervention
Gastric emptying | 240 min
Resting Energy Expenditure | At time -20 min, +60 min and +220 min

CONTACTS AND LOCATIONS:
Overall Officials: Filip K. Knop, Professor MD, Principal Investigator — Department of Clinical Medicine, University of Copenhagen, Gentofte Hospital
Locations (1):
- University Hospital, Gentofte, Copenhagen, Hellerup, Capital Region, Denmark